CLINICAL TRIAL: NCT02873455
Title: Effects of Video Information on Preoperative Anxiety in Patients With Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Heung-Kwon Oh, Clinical Associate Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1608-359-302
Record Dates: First submitted 2016-08-09; First posted 2016-08-19 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Cancer; Video Information
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- watching video (Experimental): Short video clip including the circumstance of operation theater, and surgeon's interview
  Interventions: Other: Short video clip including the circumstance of operation theater, and surgeon's interview

INTERVENTIONS:
Other: Short video clip including the circumstance of operation theater, and surgeon's interview

SUMMARY:
Patient's anxiety prior to surgery has been linked to more harmful outcome after surgery. The investigators aim to evaluate the effect of video information on preoperative anxiety level in patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-75
* Elective surgery

Exclusion Criteria:

* History of previous any surgery
* emergency surgery
* dementia
* psychological disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of APAIS ((Amsterdam preoperative anxiety and information scale) from baseline APAIS to watching video. | baseline and 1 minute after watching video.

SECONDARY OUTCOMES:
Change of HADS (Hospital Anxiety and Depression Scale) from baseline HADS to watching video. | baseline and 1 minute after watching video.
Postoperative hospital stay | through study completion and an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heung-Kwon Oh, MS, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided